CLINICAL TRIAL: NCT03663413
Title: The Oculocardiac Reflex Influenced at Different Levels of Brain Wave Monitoring
Brief Title: Oculocardiac Reflex Brain Wave Monitor
Acronym: OCRBIS
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD OCR BIS
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2018-09

CONDITIONS: Bradycardia; Strabismus
MeSH Terms: conditions — Bradycardia; Strabismus | interventions — Brain Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BIS: Monitored with BIS (bispectral index) monitor in addition to other conventional monitors of blood pressure, ECG, oxygen saturation and anesthetic agent concentration.
  Interventions: Device: non-invasive monitor
- Narcotrend: Monitored with Narcotrend monitor in addition to other conventional monitors of blood pressure, ECG, oxygen saturation and anesthetic agent concentration.
  Interventions: Device: non-invasive monitor

INTERVENTIONS:
Device: non-invasive monitor — cutaneous EEG monitor
  Other Names: brain wave

SUMMARY:
Oculocardiac reflex during routine strabismus surgery was prospectively observed in association with routine brain wave monitoring.

Providence Hospital institutional review board (IRB) approved this observational study without need for consent.

DETAILED DESCRIPTION:
Introduction: The oculocardiac reflex (OCR), bradycardia that occurs during strabismus surgery, is blocked by anticholinergics and enhanced by opioids and dexmedetomidine. Two recent studies suggest that deeper inhalational anesthesia monitored by bispectral index (BIS) protects against OCR; the investigators wondered if our data correlated similarly.

Methods: In an ongoing, prospective study of OCR elicited by 10-second, 200 gram square-wave traction on extraocular muscles (EOM) from 2009 to 2013, anesthetic depth was estimated in cohorts using either BIS or Narcotrend monitors. The depth of anesthesia was deliberately varied between first and second EOM tested.

ELIGIBILITY:
Inclusion Criteria:

* all

Exclusion Criteria:

* those receiving anticholinergic medications

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: strabismus surgery
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2009-08-27 (Actual); Primary Completion 2013-11-21 (Actual); Study Completion 2013-11-21 (Actual)

PRIMARY OUTCOMES:
heart rate change | intraoperative 10 seconds
  bradycardia with extra ocular muscle tension

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Arnold, MD, Principal Investigator — Alaska Childrens EYE & Strabismus

IPD SHARING:
Plan to Share IPD: Undecided
de-identified data base stored.

REFERENCES:
- [Background] Arnold RW, Biggs RE, Beerle BJ. Intravenous dexmedetomidine augments the oculocardiac reflex. J AAPOS. 2018 Jun;22(3):211-213.e1. doi: 10.1016/j.jaapos.2018.01.016. Epub 2018 May 5. PMID 29733898
- [Background] Arnold RW, Bond AN, McCall M, Lunoe L. The oculocardiac reflex and depth of anesthesia measured by brain wave. BMC Anesthesiol. 2019 Mar 14;19(1):36. doi: 10.1186/s12871-019-0712-z. PMID 30871507